CLINICAL TRIAL: NCT03024203
Title: A Comparison of Cognitive Training Approaches in Psychotic Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Christopher Bowie, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSYC-173-16
Record Dates: First submitted 2016-10-27; First posted 2017-01-18 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Psychotic Disorders
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Executive Training (Experimental): Executive Training (ET) involves training on computerized cognitive exercises that have graded increases in difficulty so that the participant is always challenged. A therapist will be in the room with participants to address any difficulties with the program and facilitate generation of strategies. ET will be delivered in both individual and group settings.
  Interventions: Behavioral: Cognitive Remediation - Executive Training
- Perceptual Training (Experimental): Perceptual Training (PT) involves training on computerized cognitive exercises that have graded increases in difficulty so that the participant is always challenged. A therapist will be in the room with participants to address any difficulties with the program and facilitate generation of strategies. PT will be delivered in both individual and group settings.
  Interventions: Behavioral: Cognitive Remediation - Perceptual Training

INTERVENTIONS:
Behavioral: Cognitive Remediation - Executive Training — Cognitive remediation is a cognitive and behavioural therapy designed to improve cognitive skills such as memory, and problem solving ability.
  Arms: Executive Training
Behavioral: Cognitive Remediation - Perceptual Training — Cognitive remediation is a cognitive and behavioural therapy designed to improve cognitive skills such as attention, and processing speed.
  Arms: Perceptual Training

SUMMARY:
Cognitive remediation (CR) is the best treatment to improve neurocognitive abilities for individuals with psychosis, however, there is no gold standard method of cognitive remediation available. Cognitive training refers to the training component of CR in which people practice computerized exercises that train specific cognitive abilities. There is no agreed upon approach within the field as to the type of training that is most effective with some studies, training higher level cognitive abilities, some training perceptual abilities, and others training general cognitive skills. This study will directly compare two competing methods of cognitive training on measures of neurophysiology, neurocognition, functional competence, and real-world functional performance.

ELIGIBILITY:
Inclusion Criteria:

* psychotic disorder
* No previous cognitive remediation in past 6 months

Exclusion Criteria:

* Brain injury
* Substance abuse
* Neurocognitive disorder
* Developmental Disability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change in Functional Performance - Specific Levels of Functioning (SLOF) from Baseline | Post-treatment (within 2 weeks following the end of treatment)
  Rating scale completed by participants' case managers that rates their ability to perform different everyday tasks

SECONDARY OUTCOMES:
Change in Neurocognition - MATRICS Cognitive Consensus Battery (MCCB) from Baseline | Post-treatment (within 2 weeks following the end of treatment)
  The MCCB is the gold standard cognitive assessment for schizophrenia research
Change in Neurophysiology - EEG from Baseline | Post-treatment (within 2 weeks following the end of treatment)
  Alpha and Theta band synchronization, p300, mismatch negativity
Functional Competence - Canadian Objective Assessment of Life Skills Brief (COALS-B) from Baseline | Post-treatment (within 2 weeks following the end of treatment)
  Performance based measure of real life functional skills using role-play
Change in Functional Performance - Specific Levels of Functioning (SLOF) from Baseline | Follow-Up (3 months after the end of treatment)
  Rating scale completed by participants' case managers that rates their ability to perform different everyday tasks
Change in Neurocognition - MATRICS Cognitive Consensus Battery (MCCB) from Baseline | Follow-Up (3 months after the end of treatment)
  The MCCB is the gold standard cognitive assessment for schizophrenia research
Change in Neurophysiology - EEG from Baseline | Follow-Up (3 months after the end of treatment)
  Alpha and Theta band synchronization, p300, mismatch negativity
Functional Competence - Canadian Objective Assessment of Life Skills Brief (COALS-B) from Baseline | Follow-Up (3 months after the end of treatment)
  Performance based measure of real life functional skills using role-play

CONTACTS AND LOCATIONS:
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Best MW, Milanovic M, Iftene F, Bowie CR. A Randomized Controlled Trial of Executive Functioning Training Compared With Perceptual Training for Schizophrenia Spectrum Disorders: Effects on Neurophysiology, Neurocognition, and Functioning. Am J Psychiatry. 2019 Apr 1;176(4):297-306. doi: 10.1176/appi.ajp.2018.18070849. Epub 2019 Mar 8. PMID 30845819